CLINICAL TRIAL: NCT05661071
Title: Determination of Neuropsychological Profiles of Children With Duchenne Muscular Dystrophy and Investigation of Its Effects on Motor Functions
Brief Title: Neuropsychological Profiles of Children With Duchenne Muscular Dystrophy and Its Effects on Motor Functions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Aldırmaz, Principal Investigator, Hacettepe University
Other Study IDs: GO22/310
Record Dates: First submitted 2022-12-04; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy (DMD); neuropsychological profile; cognitive status; neurodevelopmental status; motor function; balance
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Self Report

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Duchenne Muscular Dystrophy: Children with Duchenne Muscular Dystrophy (DMD) between the ages of 7 and 16 who have been diagnosed with DMD as a result of genetic testing
  Interventions: Other: Modified Mini Mental Test:; Other: The Controlled Oral Word Association Test; Other: The Central Nervous System Vital Signs; Other: Conners' Parent Rating Scale-48 (Parent Report); Other: Child Behavior Checklist 6-18 ages (Parent Report); Other: Strengths and Difficulties Questionnaire (Self-Reported); Other: Brooke Lower Extremity Functional Classification; Other: Motor Function Measurement-32 Items; Other: Four Square Step Test; Other: Six Minutes Walk Test; Other: Timed Performance Test
- Typically Developed Children: Typically Developed Children with similar physical characteristics between the ages of 7 and 16
  Interventions: Other: Modified Mini Mental Test:; Other: The Controlled Oral Word Association Test; Other: The Central Nervous System Vital Signs; Other: Conners' Parent Rating Scale-48 (Parent Report); Other: Child Behavior Checklist 6-18 ages (Parent Report); Other: Strengths and Difficulties Questionnaire (Self-Reported)

INTERVENTIONS:
Other: Modified Mini Mental Test: — To assess the cognitive function of children
Other: The Controlled Oral Word Association Test — To assess the cognitive function of children
Other: The Central Nervous System Vital Signs — To assess the cognitive function of children
Other: Conners' Parent Rating Scale-48 (Parent Report) — To assess attention-deficit/hyperactivity disorder
Other: Child Behavior Checklist 6-18 ages (Parent Report) — To assesses both child adaptive behaviors and problem behaviors.
Other: Strengths and Difficulties Questionnaire (Self-Reported) — It is a brief emotional and behavioural screening questionnaire for children and young people.
Other: Brooke Lower Extremity Functional Classification — To determine the functional status of the lower extremity
  Groups: Duchenne Muscular Dystrophy
Other: Motor Function Measurement-32 Items — To assessment of motor function and progression of weakness in neuromuscular disorders
  Groups: Duchenne Muscular Dystrophy
Other: Four Square Step Test — A test of dynamic balance and coordination that clinically assesses the participant's ability to step over objects forward, sideways, and backwards.
  Groups: Duchenne Muscular Dystrophy
Other: Six Minutes Walk Test — It evaluates the walking function and physical capacity of children at the submaximal level.
  Groups: Duchenne Muscular Dystrophy
Other: Timed Performance Test — 10 meters Walk& Run Test, Gower's(from a supine to a standing position), Right& Left Leg Standing, Ascent/Descent of 4 Steps
  Groups: Duchenne Muscular Dystrophy

SUMMARY:
This study was planned to determine neuropsychological profiles of children with Duchenne Muscular Dystrophy and investigation of its effects on motor functions & compare to typically developed peers.

DETAILED DESCRIPTION:
In this thesis, it is aimed to determine the neuropsychological profiles of children with Duchenne Muscular Dystrophy (DMD) and to investigate its effects on motor functions. The study will be carried out with children between the ages of 7 and 16 who have been diagnosed with DMD as a result of genetic testing and who applied to Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Pediatric Neuromuscular Diseases Unit for physiotherapy and rehabilitation evaluation. In addition, considering the primary purpose of the study, typically developed boys between the ages of 7 and 16 with similar physical characteristics will be included in the study and compared with children with DMD. Typically developed boys included in the study will be evaluated only with neuropsychological tests. Evaluating cognitive function from neuropsychological tests; Modified Mini Mental Test, The Controlled Oral Word Association Test,computer-based The Central Nervous System Vital Signs will be applied. To evaluate neurodevelopmental status from neuropsychological tests; Conners' Parent Rating Scale, Child Behavior Checklist, Strengths and Difficulties Questionnaire (SDQ) will be applied. To evaluate the motor functions of individuals with DMD; Brooke Lower Extremity Functional Classification, Motor Function Measurement, Four Square Step Test, Six Minutes Walk Test, Timed Performance Tests (10 meters Walk/Run Test, Gower's (from a supine to a standing position), Right/Left Leg Standing, Ascent/Descent of 4 Steps) will be used. In the study, in which the effect of the mutation region of dystrophin protein isoforms causing DMD on the neuropsychological profile of children will be investigated by comparing them with typically developed boys and the effect of this on motor function will be examined, the statistical significance level will be considered as p<0.05

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with DMD by a pediatric neurologist,
* Being between the ages of 7-16,
* Not to have any diagnosed chronic disease,
* Not having lost yet the ability to write and draw as required by neuropsychological assessments,
* Cooperate with the physiotherapist and be able to comply with their instructions.

Exclusion Criteria:

* Inability to cooperate adequately with the physiotherapist who made the evaluations,
* Have had any injury and/or surgery to the lower/upper extremities in the last 6 months, which may prevent the performance of motor function tests.

Ages: 7 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Duchenne muscular dystrophy is an X-linked disease which effects boys.
Study Population: Children with Duchenne Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Modified Mini Mental Test | only baseline
  The Mini Mental Test developed for adults was adapted to the pediatric population by making minor modifications. Test; It evaluates verbal responses including attention, orientation, memory and language skills, ability to obey verbal and written orders, write spontaneous sentences, and copy a complex drawing. The highest score that can be obtained from this test is 35, the lowest score is 0.
The Controlled Oral Word Association Test | only baseline
  This test requires the individual to name as many words as possible that begin with a given letter, i.e. K, A and S. Sixty seconds are allotted for each letter. Individuals cannot use proper names or numbers and cannot use words with different tenses or endings once the root word has been given
The Central Nervous System Vital Signs | only baseline
  Central Nervous System Vital Signs is a reimbursable assessment procedure that utilizes computerized neuropsychological tests to evaluate the neurocognitive status of patients and covers a range of mental processes from simple motor performance, attention, memory, to executive functions.
Conners' Parent Rating Scale-48 (Parent Report) | only baseline
  The Conners' Parent Rating Scale-48 contains 48 items wherein the frequency of each item is rated on a 4-point Likert scale ranging from not at all (0)-3 very much (3). The test has adequate psychometric properties and is widely used for clinical and research purposes with the attention deficit/hyperactivity disorder population
Child Behavior Checklist 6-18 ages (Parent Report) | only baseline
  The Child Behavior Checklist/6-18 assesses both child adaptive behaviors and problem behaviors. There are 112 items that assess problem behaviors and 20 items that assess adaptive behavior. Response format for problem behaviors is from 0 ("not true") to 2 ("very true"). The problem behavior items load onto two broad-band scales (Internalizing and Externalizing) and eight narrow-band scales (Rule Breaking, Aggressive Behavior, Withdrawn-Depressed, Somatic Complaints, Anxious Depressed, Social Problems, Thought Problems, and Attention Problems). The adaptive behavior items load onto three scales: Activities, Social Competence, and School Competence. A Total Competence and Total Behavior Problems score are also provided.
Strengths and Difficulties Questionnaire (Self-Reported) | only baseline
  The Strengths and Difficulties Questionnaire is a brief emotional and behavioural screening questionnaire for children and young people. The tool can capture the perspective of children. The 25 items in the test comprise 5 scales of 5 items each. The scales include: emotional symptoms subscale, conduct problems subscale, hyperactivity/inattention subscale, peer relationships problem subscale, prosocial behaviour subscale.
Brooke Lower Extremity Functional Classification | only baseline
  It was developed using the classification method based on "Vignos et al." to determine the functional status of the lower extremity. It consists of 10 different levels, ranging from Level 1 (walks independently and climbs stairs) to Level 10 (bound to bed).
Motor Function Measurement-32 Items | only baseline
  The Motor Function Measure is a scale designed for the assessment of motor function and progression of weakness in neuromuscular disorders. It is applicable to both ambulant and non-ambulant patients with a wide range of severity. The scale exists in two versions, one with 32 items for patients over 6 years of age (MFM-32), the other with 20 items for children aged from 2 to 6 years (MFM-20). Concerning the development of the scale, factor analysis identified three functional dimensions: D1 = standing position and transfers (13 items; 8 items in the short version), D2 = axial and proximal motor function (12 items; 8 in the short version), and D3 = distal motor function (7 items; 4 in the short version).
Four Square Step Test | only baseline
  It is a valid and reliable test that has been used frequently in children in recent years to evaluate dynamic balance. Sticks, each 90 cm long, are placed on the floor to form 4 squares and the squares are numbered from 1 to 4. For the test to be completed successfully, the child must quickly move from one square to the next without touching the sticks. Performance is determined by measuring the test completion time in seconds. Shorter completion time means better dynamic balance.
Six Minutes Walk Test | only baseline
  The 6-minutes walk test, which is valid and reliable for DMD patients, will evaluate the walking function and physical capacity of children at the submaximal level. The distance the child walks for 6 minutes in a 25 m corridor will be recorded in meters. A physiotherapist will walk with the children during the test and track the time with a stopwatch. The test is simple and considered an important outcome measure for children with DMD.
10 meters Walk& Run Test | only baseline
  A 10-meter distance was marked on an unobstructed, flat surface using tape. To limit the impact of acceleration and deceleration on gait speed, start and finish lines were placed 30 centimeter before and after the 10-meter distance. Participants were instructed to begin with toes on the start line and walk or run as fast as possible, without compromising safety, to the finish line.
Gower's(from a supine to a standing position) | only baseline
  Children lied down on a mat with straight position and asked them to stand up as fast as possible. Time was started when he moved and stopped when he was upright position.
Right& Left Leg Standing Test | only baseline
  Children had to maintain a one-legged stance for as long as they could with their eyes open, and allowing them to freely-move their arms. Children were verbally encouraged to maintain the one-legged standing position for as long as possible during test.
Ascent/Descent of 4 Steps | only baseline
  The children were asked to climb up the 4-step ladder with double-sided handrails as fast as possible. The time was started when his feet lifted from the ground and when both feet touched the ground, the time was stopped and recorded in seconds. After climbing the ladder, they were asked to descend as fast as possible, the time was started when the foot was lifted, and the time was stopped when both feet touched the ground and recorded in seconds.

SECONDARY OUTCOMES:
Genetic test report | only baseline
  The effect of the mutation region of dystrophin protein isoforms causing DMD on the neuropsychological profile of children will be investigated by comparing them with typically developed boys and the effect of this on motor function will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: İpek Gürbüz, Assc. Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Pediatric Neuromuscular Diseases Unit for physiotherapy and rehabilitation, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Aldirmaz E, Bulut N, Yilmaz O, Alemdaroglu-Gurbuz I. Cognitive and emotional-behavioural outcomes of Turkish Duchenne muscular dystrophy population and its association with motor function. Eur J Paediatr Neurol. 2024 Sep;52:86-94. doi: 10.1016/j.ejpn.2024.08.004. Epub 2024 Aug 18. PMID 39180809